CLINICAL TRIAL: NCT05717647
Title: Cerebral Oxygenation and Metabolism and Severe Head Injury in Paediatrics (COMetSHIP)
Acronym: COMetSHIP
Status: Active, not recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Shruti Agrawal, Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: A096238
Record Dates: First submitted 2022-05-16; First posted 2023-02-08 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric patients with severe traumatic brain injury undergoing multimodality monitoring: * Patients admitted with brain injury requiring ventilation and ICP monitoring
  * Age group: 3 years and 16 years (children under the age of three years are excluded as the triple bolt for multimodality monitoring is not currently used for this age group)
  Interventions: Other: Observational study: neuromonitoring

INTERVENTIONS:
Other: Observational study: neuromonitoring — collection of multimodality neuromonitoring data including ICP, brain tissue oxygen tension, cerebral microdialysis data

SUMMARY:
Children suffer proportionally more head injuries than any other age group and children with head injuries have the highest mortality of all children admitted with traumatic injuries. The investigators aim to investigate the factors that contribute to poor outcomes after paediatric acute brain injury by collecting observational and outcome data. Much of the brain damage that results in poor outcomes actually happens in the hours and days after the injury. This is due to several factors such as brain swelling and poor oxygen delivery to the brain. Treatment is directed to try and protect the brain against these factors. Current management of the head injured child focuses on monitoring pressure within the head. However, this does not detect all the factors that cause continuing brain damage. Special monitors that follow oxygen levels and chemical changes in the brain are used safely in adult patients but have not been widely employed in children despite their potential benefit. There is therefore the opportunity to evaluate extra monitoring of the child brain, and in doing so, help refine the management of these patients.

DETAILED DESCRIPTION:
This is an observational study evaluating changes in intracranial pressure (ICP), brain chemistry and oxygen after an acute brain injury in children. Data will be collected from ICP sensors and brain tissue oxygen sensors that are routinely used in children with severe brain injuries. In addition, microdialysis catheters, which allow chemical changes in the brain to be followed, will be used. These monitoring devices are routinely and safely used in adults with acute brain injury but have not been widely employed in children. The ICP sensor and oxygen sensor will be inserted into the head using a cranial access device. The additional chemistry monitor for this study will be inserted using the same cranial access device. The microdialysis fluid is analysed at the bedside and the resultant data is also stored electronically. The microdialysis fluid that is left over following bedside analysis will be stored and assayed further for markers of inflammation that may also be involved in brain injury.

Patients will be recruited from the Paediatric Intensive Care Unit at Addenbrooke's Hospital. The patients will have major acute brain injury requiring ventilation. Patients will be unaware of the enrolment to the study due to the nature of the brain injury and requirement of sedation. The acute phase of the study is purely observational; there is a consent waiver for acute data collection to obtain a bias free sample and ensure consecutive recruitment to be able to improve validity of the data. There is precedence of such waiver and PICUs in UK have recruited to ADAPT (Large Multinational multi-centre head injury study in children with TBI, http://www.adapttrial.org/) with consent waiver for acute phase data collection with approval from UK based ethics committee, and more recently the STARSHIP study (Studying Trends of Auto-regulation in Severe Head Injury in Paediatrics https://action.org.uk/research/improving-treatment-traumatic-brain-injuries). The investigators will ask for consent for data sharing and data use for present and future research and undertake the outcome assessments at 6 and 12 months by telephone interview. The investigators know from previous studies that families remember very little about what was told soon after the injury and are therefore not able to provide valid informed consent. The investigators will wait until the child's condition is stable and the family has had a chance to get acclimatized to hospital and the extent of the child's injuries. At a time when the child's condition has stabilized and recovery has begun, the site PI (or a designated member of the research team) will approach the family or the person with parental responsibility to seek written informed consent. In all cases as far as possible, consent will be obtained prior to hospital discharge.

Mortality at 30 days and at 12 months will be evaluated as a primary outcome measure. Functional outcomes will be evaluated at 6 and 12 months when patients are routinely seen for clinical follow--up. Outcomes will be assessed using the Pediatric Quality of Life Inventory (PedsQL) and the Glasgow Outcome Scale - Extended Pediatric Revision (GOS--E Peds) by asking the parent/guardian to complete the relevant questionnaires during the clinic appointment or to return the questionnaire by post after the appointment. Comparison between ICP, brain tissue oxygen and microdialysis results will be made by calculating median values, interquartile ranges, confidence intervals and by using non-parametric statistical hypothesis tests (Man--Whitney U/ Wilcoxon signed--rank test). It is noted that this is an observational study and data collected will not guide treatment.

Given the critical condition of the brain injured patients recruited to this study there is an expectation that a proportion of participants will die despite treatment, and that the survivors will have a range of neurological deficits, that may be highly disabling. Furthermore, adverse events (e.g. sepsis) are common in this patient group. Reflecting this, an extended period of treatment in the Paediatric Intensive Care Unit and as a ward inpatient is likely. Therefore the investigators will record and report adverse events relevant to the study procedures and any serious adverse events that are related or potentially related to the study procedures.

Study sample data will be anonymised and coded using a study identifier. Anonymised research data will be stored on computers within the Division of Neurosurgery in an encrypted password-protected format. No one outside the direct study team will have access to this data. The Principal and Lead investigators will ultimately be responsible for storing all data (electronic and paper) securely in compliance with The Data Protection Act 1998.

The study is to be carried out in conformation with the spirit and the letter of the declaration of Helsinki, and in accord with the ICH Good Clinical Practice Guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with brain injury requiring ventilation and ICP monitoring
* Age group: 3 years and 16 years (children under the age of three years are excluded as the triple bolt for multimodality monitoring is not currently used for this age group)

Exclusion Criteria:

* Bleeding diathesis
* Patient unlikely to survive more than 24 hours

Ages: 3 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Paediatric patients with severe brain injury undergoing multimodality neuromonitoring
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  Death at 30 days
Mortality | 12 months
  Death at 12 months

SECONDARY OUTCOMES:
PedsQL | 6 and 12 months
  Assessed using the Pediatric Quality of Life Inventory
  minimum score = 0 maximum score = 100 higher score indicates a better outcome
Functional outcomes | 6 and 12 months
  Assessed using the Glasgow Outcome Scale - Extended Pediatric Revision
  minimum value = 1 maximum value = 8 higher value indicates a worse outcome
Correlation of lactate to pyruvate ratio (LPR) with intracranial pressure, cerebral perfusion pressure and brain tissue oxygenation | End of Neuro-monitoring period (upto 2 weeks)
  LPR values are indicative of the anaerobic metabolism and substrate deliver. From adult studies, LPR >25 is considered abnormal. The investigators will be assessing LPR values with the other neuro-monitoring variables as described above to assess whether the same values are applicable in children.
  There will be LPR readings every hour from microdialysis samples.
Functional outcomes in relation to LPR | 6 and 12 months
  Correlation of LPR with functional outcomes as assessed by Glasgow Outcome Scale- Extended Pediatric and Pediatric Quality of Life Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Agrawal, Principal Investigator — Shruti Agrawal
Locations (1):
- Cambridge University Hospitals, Cambridge, Cambridgeshire, United Kingdom